CLINICAL TRIAL: NCT04033536
Title: A Prospective Randomized Trial of Involved Versus Elective Target Definition in Stereotactic Spine Radiosurgery for Spinal Metastases
Brief Title: Involved Versus Elective Target SSRS for Spinal Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201905015RINC
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Secondary Malignant Neoplasm of Spine
Keywords: Spine metastasis; Stereotactic spine radiosurgery; Target definition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Involved target SSRS (Active Comparator): Spine stereotactic radiosurgery/ablative radiotherapy (SSRS) with 16 Gy in single fraction to the defined Involved Target Volume using intensity modulated radiotherapy or volumetric modulated arc therapy (VMAT or RapidArc).
  Interventions: Radiation: Involved Target Stereotacic Spine Radiosurgery
- Elective target SSRS (Active Comparator): SSRS with 16 Gy in single fraction to the defined Elective Target Volume using intensity modulated radiotherapy or volumetric modulated arc therapy (VMAT or RapidArc).
  Interventions: Radiation: Elective Target Stereotacic Spine Radiosurgery

INTERVENTIONS:
Radiation: Involved Target Stereotacic Spine Radiosurgery — Image guidance spine stereotactic radiosurgery/ablative radiotherapy 1600 cGy in single fraction to Involved Target using IMRT/VMAT/RapidArc
  Arms: Involved target SSRS
Radiation: Elective Target Stereotacic Spine Radiosurgery — Image guidance spine stereotactic radiosurgery/ablative radiotherapy 1600 cGy in single fraction to Elective Target using IMRT/VMAT/RapidArc
  Arms: Elective target SSRS

SUMMARY:
The spine is a common metastatic site for malignancy and it can lead to serious and devastating events, including pain, neurological dysfunction, and reduction in quality of life. The radiotherapy (RT) has been the mainstay for palliating painful spinal metastases for the past decades. It is utilized to arrest the tumor growth, control pain, and stabilize or improve skeletal and/or neurological function. One of the limitations of the conventional radiotherapy is that radiation dose intensification is not achievable with conventional RT techniques due to the dose-limiting spinal cord, which is close to the vertebral body and sometimes encased by epidural lesion.

The management of patients with spine metastasis has undergone a great deal of change in the past 10 years. The concept of radiosurgery, a high dose of radiation targeted to a pathological entity and delivered in 1-5-fractions, has proven so successful at treating both benign and malignant lesions that it changed the paradigm for radiation therapy. Clinical experiences with high dose spine stereotactic radiosurgery (SSRS) for spinal metastases demonstrated both safety and efficacy. Nontheless, the patterns of clinical practice of SSRS varies considerably regarding the dose fractionation, target delineation, and dosimetry. There is lack of evidence-based recommedations for SSRS.

In our prior clinical trial comparing single fraction and multiple fractions SSRS (NCT02608866), single-fraction with 16 Gy is the preferred regimen for further evaluation since it met the predefined primary endpoint and has lower risk of treatment failure compared to the multiple-fraction arm. Regarding the target volume definition, the International Spine Radiosurgery Consortium published concensus guidelines based on expert opinions and limited case series. We proposed this randomized study to determine the preferred or acceptable definition of target volume delineation in SSRS and to evaluate their toxicity, efficacy, and patterns of failure. Our analysis will provide evidence-based recommendations as well as predictive factors regarding the clinical practice of SSRS.

DETAILED DESCRIPTION:
Although conventionally fractionated radiation therapy has been utilized for decades, the rates of complete pain relief and local control for complex tumors are sub-optimal. The management of patients with spine metastasis has undergone a great deal of change in the past 5 years. Improvements in neuroimaging, computer- assited treatment planning, and radiation therapy techniques have led to the development of extracranial radiosurgery.

SSRS is rapidly being adopted in the clinic as preliminary applications of SSRS appears promising. However, the role of SSRS remains in its infancy and lacked high-quality evidence about the treatment schedule and lacked a solid understanding of the adverse events. The RTOG 0631 phase 2/3 study was initiated to determine whether a more intensive radiation dose delivered by image guided 16-Gy dose single fraction SRS could improve pain control and quality of life as compared with conventional EBRT in patients with localized spine metastases. Our preliminary result from previus phase 2 stereotactic spine radiosurgery trial (NCT02608866) also showed good local control with minimal side effects in the single fraction 16-Gy setting as compared with 3 fractions 24 -Gy SRS dose.

Accurate and approproate delineation of the target area is paramount to the utilization of spine SBRT. Whethr the target volume should include the entire extent of tumor and the involved anatomical compartment for intact vertebra metastasis or remained to be discussed.

Our preliminary showed that the overall treatment failure rate was only about 14% using the definition of the treating the affected spinal lesions(invovled target ) instead of treating the entire . Better dose coverage of the target vome with improved normal tissue protection can be achived with invovled field treatment without compromising the local control. Since no treamtent target consensus has been reached from current clinical practive evidence. It is pivotal to establish and collect more treatment evidence for future spinal SBRT.

There was no randomized trials to assess the SSRS treatment response and SSRS induced grade 3 or higher adverse events between these two different target delineations. Thus, we proposed the randomized study to determine the feasibility of using "Invovled Target Volume" versus "Elective Target Volume" and tried to evaluate the toxicity profile and gain robust data as well as predictive factors regarding the local control rate and risk of complications after SSRS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of non-hematopoietic malignancy
* Radiographic evidence of localized spine metastases without leptomeningeal involvement or intramedullary lesion
* Maximum four separate sites with a maximal involvement of two continuous vertebral levels
* Patients do not have prior radiotherapy to the index spine(s)
* Age ≥ 20 years
* Karnofsky performance status (KPS) ≥ 60%.
* Life expectancy of ≥ 6 month.
* Women of childbearing potential and male participants must practice adequate contraception
* Patients must be able to comply with the study protocol and follow- up schedules and provide study-specific informed consent

Exclusion Criteria:

* Prior radiotherapy to the index spine(s)
* Serum creatinine > 2.0 mg/dL within 90 days prior registration
* Contraindication to MR imaging such as implanted metal devices or foreign bodies, severe claustrophobia
* Patients with leptomeningeal involvement or intramedullary metastasis
* Inability to tolerate treatment procedure
* Bony retropulsion causing neurologic abnormality
* Severe, active comorbidities which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the protocol, or limit compliance with study requirements
* Will receive any other investigational agent or chemotherapy and/or target therapies during treatment
* Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study may be significantly teratogenic
* Pregnant or breast-feeding women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Treatment Failure Rate at 6 months after SSRS | 6 months
  The rate of predefined treatment failure at 6-month after stereotactic spine radiosurgery. Treatment failure is defined as Grade 3 or higher adverse events definitely, probably, or possibly related to treatment and/or unequivocal local progression indicative of surgical intervention or re-irradiation.

SECONDARY OUTCOMES:
Health-related quality of life for palliative cancer care | 1-, 3-, and 6-month, and every 3 months thereafter until neurological progression, death, or up to 1 year after SSRS
  EORTC QLQ-C15-PAL Taiwan

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Ming Hsu, M.D., Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No